CLINICAL TRIAL: NCT06520683
Title: Short-course PD-1 Blockade As Adjuvant Treatment for High-risk Stage-II DMMR/MSI-H Colorectal Cancer
Brief Title: Adjuvant PD-1 Blockade for High-risk Stage-II DMMR/MSI-H Colorectal Cancer
Acronym: SMALLER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Pei-Rong Ding, Director of the Department of Colorectal Surgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-219
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Microsatellite Instability High
Keywords: Adjuvant therapy; Stage II CRC; dMMR/MSI-H; PD-1 blockade
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tislelizumab Arm (Experimental): Two cycles of Tislelizumab 200mg intravenously, on day 1 and day 22, with or without adjuvant chemotherapy
  Interventions: Drug: Tislelizumab; Drug: Adjuvant chemotherapy
- Control Arm (Active Comparator): Receiving standard of Care (either with adjuvant chemotherapy or surveillance alone).
  Interventions: Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Tislelizumab — - Tislelizumab 200mg (day 1 and day 22), administered after surgery
  Other Names: Tislelizumab (Tevimbra)
  Arms: Tislelizumab Arm
Drug: Adjuvant chemotherapy — * Adjuvant therapy is not mandatory.
  * Optional adjuvant regimens include FOLFOX, CapeOX, 5-FU+LV, or Capecitabine.

SUMMARY:
This open-label phase III trial investigates the efficacy of two cycles of PD-1 blockade (Tislelizumab) as adjuvant therapy to see how it works compared with standard of care (SOC) in treating patients with stage II dMMR/MSI-H colorectal cancer.

The rational of giving PD-1 blockade as adjuvant therapy is based on the fact that tumor recurrence is extremely low among patients receiving neoadjuvant immunotherapy, which suggests that PD-1 blockade may likely improve patients' long-term survival.

As for the short course (two cycles), we have the following considerations: firstly, the NICHE-2 trial, which adopted a two-cycle regimen, reported no recurrences during follow-up, suggesting that short-course anti-PD-1 therapy may be sufficient to improve the survival of patients with localized dMMR/MSI-H colorectal cancer. Secondly, the potential benefits of PD-1 blockade should be balanced against its toxicities, because patients with stage-II dMMR colorectal cancer generally have a good prognosis. Two cycles of PD-1 blockade have been shown to have a good safety profile, with low incidence of grade 3-4 and immune-related adverse events.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, randomised, phase III trial comparing the combination of PD-1 blockade + SOC versus SOC alone as adjuvant therapy for patients with high-risk stage-II dMMR/MSI-H colorectal cancer.

Primary Objective: To determine whether the addition of Tislelizumab can significantly improve disease-free survival (DFS) compared to standard of care in patients with high-risk stage-II colorectal cancer.

Secondary objectives:

* To determine whether the addition of Tislelizumab can significantly improve overall survival (OS) compared to standard of care
* To assess the adverse events (AE) profile (including immune-related adverse events, ir-AEs).

OUTLINE: Patients are randomized to 1 of 2 arms, stratified by cT4 status.

Arm 1 (experimental group): patients receive Tislelizumab 200mg intravenously on day 1, with or without adjuvant chemotherapy, and repeat the treatment on day 22. Patients undergo routine follow-up every 3 months for the first 3 years, and then every 6 months for the year 4-5.

Arm 2 (control group): patients receive standard of care (SOC), whether with surveillance alone, single-agent Capecitabine, or CapeOx/FOLFOX, at the discretion of the doctor in charge. Patients undergo routine follow-up every 3 months for the first 3 years, and then every 6 months for the year 4-5.

Statistics According to the statistical design, 180 patients (90 per arm) are to be randomized. The study is expected to take up to 36 months to complete accrual.

ELIGIBILITY:
Inclusion Criteria:

* dMMR and/or MSI-H colorectal carcinoma that undergo surgical resection
* Pathologically confirmed as stage II (T3-4,N0), with at least one of the following risk factors: 1) T4 (including T4a and T4b); 2) Vascular invasion; 3) Perineural invasion; 4) Poor differentiation (including mucinous and signet-ring carcinoma); 5) Obstruction and/or perforation before surgery.
* Perioperative CT/MR/PET-CT find no signs of metastases
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days prior to study start
* Aged 18-80
* No prior medical therapy (chemotherapy, immunotherapy, biologic or targeted therapy) or radiation therapy for the current cancer
* Adequate organ function

Exclusion Criteria:

* Active autoimmune disease that has required systemic treatment in past 2 years
* Positive surgical margin (R1/R2 resection)
* Presence of post-operative complications that may preclude treatment
* Active infection requiring systemic therapy
* Any other malignant disease within the preceding 5 years with the exception of non-melanomatous skin cancer, carcinoma in situ and early stage disease with a recurrence risk <5%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  DFS (tumor-specific) is defined as time from randomization to tumor relapse or tumor-related death. DFS will be compared between treatment arms using the stratified log rank test at one-sided level 0.025. If zero DFS events are observed in a certain stratum at an interim analysis and unstratified log-rank is used, all subsequent analyses for DFS will use unstratified log-rank test.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  OS is defined as time from randomization to death from any cause. Overall survival will be compared between treatment arms using the log-rank test.
Incidence of adverse events | up to 30 days after last treatment
  Assessed by Common Terminology Criteria for Adverse Events version 4.0. The overall adverse event rates and the immune-related adverse event rates will be compared between treatment arms using Chi-square test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Rong Ding, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Dept. of Colorectal Surgery, Sun Yat-sen University Cancer Center. Yuexiu District, Dongfeng East Road 651, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No